CLINICAL TRIAL: NCT01174550
Title: PROspective Multicenter Imaging Study for Evaluation of Chest Pain - The PROMISE Trial
Brief Title: PROspective Multicenter Imaging Study for Evaluation of Chest Pain
Acronym: PROMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00019865; R01HL098237-01 (NIH)
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Chest Pain
Keywords: chest pain; coronary artery disease; CAD
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional diagnostic tests (Active Comparator): Stress Echocardiogram Nuclear Stress Test Exercise Electrocardiogram
  Interventions: Procedure: Stress Echocardiogram; Procedure: Nuclear Stress Test; Procedure: Exercise Electrocardiogram
- Anatomic diagnostic test (Active Comparator): Coronary Angiography
  Interventions: Procedure: Coronary Angiography

INTERVENTIONS:
Procedure: Coronary Angiography — Use of standard equipment for usual-care testing
  Arms: Anatomic diagnostic test
Procedure: Stress Echocardiogram — Use of standard equipment for usual-care testing
  Arms: Functional diagnostic tests
Procedure: Nuclear Stress Test — Use of standard equipment for usual-care testing
  Arms: Functional diagnostic tests
Procedure: Exercise Electrocardiogram — Use of standard equipment for usual-care testing
  Arms: Functional diagnostic tests

SUMMARY:
A prospective multicenter imaging study for evaluation of chest pain. Objective is to determine whether an initial non-invasive anatomic imaging strategy with coronary CT angiography (CTA) will improve clinical outcomes in subjects with symptoms concerning for coronary artery disease relative to an initial functional testing strategy (usual care). Study hypothesis: initial anatomic testing strategy will provide information that will result in superior long-term health outcomes as compared to an initial functional testing strategy.

DETAILED DESCRIPTION:
Pragmatic randomized trial of clinical effectiveness of diagnostic testing strategies for coronary artery disease (CAD), to be performed in outpatient settings including acute and primary care and cardiology offices. Qualifying patients presenting with new or worsening symptoms suspicious for clinically significant CAD who require diagnostic testing and have not been previously evaluated will be randomized to an initial strategy of either anatomic or functional testing. All subsequent decisions regarding additional testing, medications and/or procedures will be at the discretion of the responsible clinical care team Within the functional testing arm, the subject's care team will select the specific test to be performed (exercise electrocardiogram (ECG), stress nuclear, or stress echocardiogram (echo)) consistent with 'usual care' in that practice setting. The subject's care team will be provided with 'Information sheets' summarizing current standards for test interpretation and preventive care, but specific medical treatment will not be mandated by the trial.

ELIGIBILITY:
Inclusion Criteria:

* new or worsening chest pain suspicious for clinically significant coronary artery disease (CAD)
* no prior evaluation for this episode of symptoms
* planned non-invasive testing for diagnosis
* men age ≥55 years
* men age ≥45 years with increased probability of coronary artery disease (CAD) due to either (A. Diabetes Mellitus (DM) requiring medical treatment OR Peripheral Arterial Disease (PAD) defined as documented >50% peripheral arterial stenosis treated medically or invasively OR cerebrovascular disease (stroke, documented > 50% carotid stenosis treated medically or invasively) OR B. At least one of the following cardiovascular risk factors: 1-Ongoing tobacco use, 2-Hypertension, 3-Abnormal ankle brachial index (ABI) defined as less than <0.9, 4-Dyslipidemia
* women age ≥65 years
* women age ≥50 years with increased probability of coronary artery disease (CAD) due to either (A. Diabetes Mellitus (DM) requiring medical treatment OR Peripheral Arterial Disease (PAD) defined as documented >50% peripheral arterial stenosis treated medically or invasively OR cerebrovascular disease (stroke, documented > 50% carotid stenosis treated medically or invasively) OR B. At least one of the following cardiovascular risk factors: 1-Ongoing tobacco use, 2-Hypertension, 3-Abnormal ankle brachial index (ABI) defined as less than <0.9, 4-Dyslipidemia
* Serum creatinine ≤ 1.5 mg/dL within the past 90 days
* Negative urine/serum pregnancy test for female subjects of child-bearing potential

Exclusion Criteria:

* Diagnosed or suspected acute coronary syndrome (ACS) requiring hospitalization or urgent or emergent testing; Elevated troponin or creatine kinase-myocardial band (CK-MB)
* Hemodynamically or clinically unstable condition systolic blood pressure (BP) < 90 mmHg, atrial or ventricular arrhythmias, or persistent resting chest pain felt to be ischemic despite adequate therapy)
* Known coronary artery disease (CAD) with prior Myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or any angiographic evidence of coronary artery disease (CAD) ≥50% lesion in a major epicardial vessel
* Any invasive coronary angiography or non-invasive anatomic or functional cardiovascular (CV) test for detection of coronary artery disease (CAD), including coronary tomographic angiography (CTA) and exercise electrocardiogram (ECG), within the previous twelve (12) months
* Known significant congenital, valvular (> moderate) or cardiomyopathic process (hypertrophic cardiomyopathy or reduced systolic left ventricular function (LVEF) ≤ 40%)) which could explain cardiac symptoms
* Contraindication to undergoing a coronary tomographic angiography (CTA), including but not limited to: a. Allergy to iodinated contrast agent, b. Unable to receive beta blockers unless heart rate < 65 beats per minute, c. Pregnancy
* Life expectancy < 2 years
* Unable to provide written informed consent or participate in long-term follow-up

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10003 (Actual)
Dates: Start 2010-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela S Douglas, MD, Principal Investigator — Duke Clinical Research Institute
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted to the NHLBI according to their guidelines which state"The data sets must be submitted to the study NHLBI study Program Official no later than 3 years after the end of the clinical activity (final patient follow-up, etc.) or 2 years after the main paper of the trial has been published, whichever comes first. Data are prepared by the study coordinating center and sent to the PO for review prior to release."

REFERENCES:
- [Derived] Karady J, Mayrhofer T, Brendel JM, Kolossvary M, Langenbach M, Langenbach I, Baliyan V, Sturniolo AK, Pagidipati N, Lu MT, Ferencik M, Shah S, Douglas PS, Foldyna B. Prognostic Value of Plaque Volume in Patients With First Diagnosis of Coronary Artery Disease: A Substudy of the PROMISE Randomized Clinical Trial. JAMA Cardiol. 2026 Feb 11. doi: 10.1001/jamacardio.2025.5520. Online ahead of print. PMID 41670958
- [Derived] Douglas PS, Stebbins A, Foldyna B, Patel MR, Mark DB, Lu MT, Hoffmann U, Shah SH, Martinez B, Alhanti B, Pagidipati N. Survival After Initial Stress Testing vs Anatomic Testing in Suspected Coronary Artery Disease: Long-Term Follow-Up of the PROMISE Randomized Clinical Trial. JAMA Cardiol. 2025 Oct 1;10(10):1050-1054. doi: 10.1001/jamacardio.2025.2882. PMID 40864459
- [Derived] Rasmussen LD, Sikjaer M, Soby JH, Pedersen OB, Westra J, Efthekhari A, Christiansen EH, Foldyna B, Williams MC, Dweck MR, Newby DE, Douglas PS, Bottcher M, Winther S. Dual probability approach for risk adjustment in patients with a low clinical likelihood of coronary artery disease. Eur Heart J Cardiovasc Imaging. 2025 Aug 29;26(9):1507-1517. doi: 10.1093/ehjci/jeaf193. PMID 40590244
- [Derived] McGarrah RW, Ferencik M, Giamberardino SN, Hoffmann U, Foldyna B, Karady J, Ginsburg GS, Kraus WE, Douglas PS, Shah SH. Lipoprotein Subclasses Associated With High-Risk Coronary Atherosclerotic Plaque: Insights From the PROMISE Clinical Trial. J Am Heart Assoc. 2023 Jan 3;12(1):e026662. doi: 10.1161/JAHA.122.026662. Epub 2022 Dec 24. PMID 36565187
- [Derived] Karady J, Ferencik M, Mayrhofer T, Meyersohn NM, Bittner DO, Staziaki PV, Szilveszter B, Hallett TR, Lu MT, Puchner SB, Simon TG, Foldyna B, Ginsburg GS, McGarrah RW, Voora D, Shah SH, Douglas PS, Hoffmann U, Corey KE. Risk factors for cardiovascular disease among individuals with hepatic steatosis. Hepatol Commun. 2022 Dec;6(12):3406-3420. doi: 10.1002/hep4.2090. Epub 2022 Oct 25. PMID 36281983
- [Derived] Ferencik M, Mayrhofer T, Lu MT, Bittner DO, Emami H, Puchner SB, Meyersohn NM, Ivanov AV, Adami EC, Voora D, Ginsburg GS, Januzzi JL, Douglas PS, Hoffmann U. Coronary Atherosclerosis, Cardiac Troponin, and Interleukin-6 in Patients With Chest Pain: The PROMISE Trial Results. JACC Cardiovasc Imaging. 2022 Aug;15(8):1427-1438. doi: 10.1016/j.jcmg.2022.03.016. Epub 2022 May 11. PMID 35926901
- [Derived] Lowenstern A, Alexander KP, Pagidipati NJ, Hill CL, Pellikka PA, Cooper LS, Alhanti B, Hoffmann U, Mark DB, Douglas PS. Presenting Symptoms in Patients Undergoing Coronary Artery Disease Evaluation: Association With Noninvasive Test Results and Clinical Outcomes in the PROMISE Trial. Circ Cardiovasc Qual Outcomes. 2022 May;15(5):e008298. doi: 10.1161/CIRCOUTCOMES.121.008298. Epub 2022 Apr 4. PMID 35369715
- [Derived] Fordyce CB, Hill CL, Mark DB, Alhanti B, Pellikka PA, Hoffmann U, Patel MR, Douglas PS; PROMISE Investigators. Physician judgement in predicting obstructive coronary artery disease and adverse events in chest pain patients. Heart. 2022 May 12;108(11):860-867. doi: 10.1136/heartjnl-2021-320275. PMID 35110385
- [Derived] Kammerlander AA, Mayrhofer T, Ferencik M, Pagidipati NJ, Karady J, Ginsburg GS, Lu MT, Bittner DO, Puchner SB, Bihlmeyer NA, Meyersohn NM, Emami H, Shah SH, Douglas PS, Hoffmann U; PROMISE Investigators. Association of Metabolic Phenotypes With Coronary Artery Disease and Cardiovascular Events in Patients With Stable Chest Pain. Diabetes Care. 2021 Apr;44(4):1038-1045. doi: 10.2337/dc20-1760. Epub 2021 Feb 8. PMID 33558267
- [Derived] Meyersohn NM, Mayrhofer T, Corey KE, Bittner DO, Staziaki PV, Szilveszter B, Hallett T, Lu MT, Puchner SB, Simon TG, Foldyna B, Voora D, Ginsburg GS, Douglas PS, Hoffmann U, Ferencik M. Association of Hepatic Steatosis With Major Adverse Cardiovascular Events, Independent of Coronary Artery Disease. Clin Gastroenterol Hepatol. 2021 Jul;19(7):1480-1488.e14. doi: 10.1016/j.cgh.2020.07.030. Epub 2020 Jul 21. PMID 32707340
- [Derived] Goyal A, Pagidipati N, Hill CL, Alhanti B, Udelson JE, Picard MH, Pellikka PA, Hoffmann U, Mark DB, Douglas PS. Clinical and Economic Implications of Inconclusive Noninvasive Test Results in Stable Patients With Suspected Coronary Artery Disease: Insights From the PROMISE Trial. Circ Cardiovasc Imaging. 2020 Apr;13(4):e009986. doi: 10.1161/CIRCIMAGING.119.009986. Epub 2020 Apr 9. PMID 32268807
- [Derived] Lowenstern A, Alexander KP, Hill CL, Alhanti B, Pellikka PA, Nanna MG, Mehta RH, Cooper LS, Bullock-Palmer RP, Hoffmann U, Douglas PS. Age-Related Differences in the Noninvasive Evaluation for Possible Coronary Artery Disease: Insights From the Prospective Multicenter Imaging Study for Evaluation of Chest Pain (PROMISE) Trial. JAMA Cardiol. 2020 Feb 1;5(2):193-201. doi: 10.1001/jamacardio.2019.4973. PMID 31738382
- [Derived] Litwin SE, Coles A, Hill CL, Alhanti B, Pagidipati N, Lee KL, Pellikka PA, Mark DB, Udelson JE, Cooper L, Tardif JC, Hoffmann U, Douglas PS; PROMISE investigators. Discordances between predicted and actual risk in obese patients with suspected cardiac ischaemia. Heart. 2020 Feb;106(4):273-279. doi: 10.1136/heartjnl-2018-314503. Epub 2019 Oct 10. PMID 31601728
- [Derived] Litwin SE, Coles A, Pagidipati N, Lee KL, Pellikka PA, Mark DB, Udelson JE, Hoffmann U, Douglas PS; PROMISE Investigators. Effects of obesity on noninvasive test results in patients with suspected cardiac ischemia: Insights from the PROMISE trial. J Cardiovasc Comput Tomogr. 2019 Jul-Aug;13(4):211-218. doi: 10.1016/j.jcct.2019.03.010. Epub 2019 Mar 27. PMID 30954400
- [Derived] Sharma A, Coles A, Sekaran NK, Pagidipati NJ, Lu MT, Mark DB, Lee KL, Al-Khalidi HR, Hoffmann U, Douglas PS. Stress Testing Versus CT Angiography in Patients With Diabetes and Suspected Coronary Artery Disease. J Am Coll Cardiol. 2019 Mar 5;73(8):893-902. doi: 10.1016/j.jacc.2018.11.056. PMID 30819356
- [Derived] Jang JJ, Bhapkar M, Coles A, Vemulapalli S, Fordyce CB, Lee KL, Udelson JE, Hoffmann U, Tardif JC, Jones WS, Mark DB, Sorrell VL, Espinoza A, Douglas PS, Patel MR; PROMISE Investigators. Predictive Model for High-Risk Coronary Artery Disease. Circ Cardiovasc Imaging. 2019 Feb;12(2):e007940. doi: 10.1161/CIRCIMAGING.118.007940. PMID 30712364
- [Derived] Januzzi JL Jr, Suchindran S, Hoffmann U, Patel MR, Ferencik M, Coles A, Tardif JC, Ginsburg GS, Douglas PS; PROMISE Investigators. Single-Molecule hsTnI and Short-Term Risk in Stable Patients With Chest Pain. J Am Coll Cardiol. 2019 Jan 29;73(3):251-260. doi: 10.1016/j.jacc.2018.10.065. PMID 30678753
- [Derived] Pagidipati NJ, Coles A, Hemal K, Lee KL, Dolor RJ, Pellikka PA, Mark DB, Patel MR, Litwin SE, Daubert MA, Shah SH, Hoffmann U, Douglas PS; PROMISE Investigators. Sex differences in management and outcomes of patients with stable symptoms suggestive of coronary artery disease: Insights from the PROMISE trial. Am Heart J. 2019 Feb;208:28-36. doi: 10.1016/j.ahj.2018.11.002. Epub 2018 Nov 9. PMID 30529930
- [Derived] Adamson PD, Newby DE, Hill CL, Coles A, Douglas PS, Fordyce CB. Comparison of International Guidelines for Assessment of Suspected Stable Angina: Insights From the PROMISE and SCOT-HEART. JACC Cardiovasc Imaging. 2018 Sep;11(9):1301-1310. doi: 10.1016/j.jcmg.2018.06.021. PMID 30190030
- [Derived] Januzzi JL Jr, Suchindran S, Coles A, Ferencik M, Patel MR, Hoffmann U, Ginsburg GS, Douglas PS; PROMISE Investigators. High-Sensitivity Troponin I and Coronary Computed Tomography in Symptomatic Outpatients With Suspected CAD: Insights From the PROMISE Trial. JACC Cardiovasc Imaging. 2019 Jun;12(6):1047-1055. doi: 10.1016/j.jcmg.2018.01.021. Epub 2018 Mar 14. PMID 29550314
- [Derived] Ferencik M, Mayrhofer T, Bittner DO, Emami H, Puchner SB, Lu MT, Meyersohn NM, Ivanov AV, Adami EC, Patel MR, Mark DB, Udelson JE, Lee KL, Douglas PS, Hoffmann U. Use of High-Risk Coronary Atherosclerotic Plaque Detection for Risk Stratification of Patients With Stable Chest Pain: A Secondary Analysis of the PROMISE Randomized Clinical Trial. JAMA Cardiol. 2018 Feb 1;3(2):144-152. doi: 10.1001/jamacardio.2017.4973. PMID 29322167
- [Derived] Lu MT, Meyersohn NM, Mayrhofer T, Bittner DO, Emami H, Puchner SB, Foldyna B, Mueller ME, Hearne S, Yang C, Achenbach S, Truong QA, Ghoshhajra BB, Patel MR, Ferencik M, Douglas PS, Hoffmann U. Central Core Laboratory versus Site Interpretation of Coronary CT Angiography: Agreement and Association with Cardiovascular Events in the PROMISE Trial. Radiology. 2018 Apr;287(1):87-95. doi: 10.1148/radiol.2017172181. Epub 2017 Nov 27. PMID 29178815
- [Derived] Sharma A, Sekaran NK, Coles A, Pagidipati NJ, Hoffmann U, Mark DB, Lee KL, Al-Khalidi HR, Lu MT, Pellikka PA, Truong QA, Douglas PS. Impact of Diabetes Mellitus on the Evaluation of Stable Chest Pain Patients: Insights From the PROMISE (Prospective Multicenter Imaging Study for Evaluation of Chest Pain) Trial. J Am Heart Assoc. 2017 Oct 31;6(11):e007019. doi: 10.1161/JAHA.117.007019. PMID 29089344
- [Derived] Ladapo JA, Coles A, Dolor RJ, Mark DB, Cooper L, Lee KL, Goldberg J, Shapiro MD, Hoffmann U, Douglas PS. Quantifying sociodemographic and income disparities in medical therapy and lifestyle among symptomatic patients with suspected coronary artery disease: a cross-sectional study in North America. BMJ Open. 2017 Sep 29;7(9):e016364. doi: 10.1136/bmjopen-2017-016364. PMID 28965093
- [Derived] Budoff MJ, Mayrhofer T, Ferencik M, Bittner D, Lee KL, Lu MT, Coles A, Jang J, Krishnam M, Douglas PS, Hoffmann U; PROMISE Investigators. Prognostic Value of Coronary Artery Calcium in the PROMISE Study (Prospective Multicenter Imaging Study for Evaluation of Chest Pain). Circulation. 2017 Nov 21;136(21):1993-2005. doi: 10.1161/CIRCULATIONAHA.117.030578. Epub 2017 Aug 28. PMID 28847895
- [Derived] Lu MT, Douglas PS, Udelson JE, Adami E, Ghoshhajra BB, Picard MH, Roberts R, Lee KL, Einstein AJ, Mark DB, Velazquez EJ, Carter W, Ridner M, Al-Khalidi HR, Hoffmann U. Safety of coronary CT angiography and functional testing for stable chest pain in the PROMISE trial: A randomized comparison of test complications, incidental findings, and radiation dose. J Cardiovasc Comput Tomogr. 2017 Sep-Oct;11(5):373-382. doi: 10.1016/j.jcct.2017.08.005. Epub 2017 Aug 15. PMID 28838846
- [Derived] Hoffmann U, Ferencik M, Udelson JE, Picard MH, Truong QA, Patel MR, Huang M, Pencina M, Mark DB, Heitner JF, Fordyce CB, Pellikka PA, Tardif JC, Budoff M, Nahhas G, Chow B, Kosinski AS, Lee KL, Douglas PS; PROMISE Investigators. Prognostic Value of Noninvasive Cardiovascular Testing in Patients With Stable Chest Pain: Insights From the PROMISE Trial (Prospective Multicenter Imaging Study for Evaluation of Chest Pain). Circulation. 2017 Jun 13;135(24):2320-2332. doi: 10.1161/CIRCULATIONAHA.116.024360. Epub 2017 Apr 7. PMID 28389572
- [Derived] Fordyce CB, Douglas PS, Roberts RS, Hoffmann U, Al-Khalidi HR, Patel MR, Granger CB, Kostis J, Mark DB, Lee KL, Udelson JE; Prospective Multicenter Imaging Study for Evaluation of Chest Pain (PROMISE) Investigators. Identification of Patients With Stable Chest Pain Deriving Minimal Value From Noninvasive Testing: The PROMISE Minimal-Risk Tool, A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2017 Apr 1;2(4):400-408. doi: 10.1001/jamacardio.2016.5501. PMID 28199464
- [Derived] Ladapo JA, Hoffmann U, Lee KL, Coles A, Huang M, Mark DB, Dolor RJ, Pelberg RA, Budoff M, Sigurdsson G, Severance HW, Douglas PS. Changes in Medical Therapy and Lifestyle After Anatomical or Functional Testing for Coronary Artery Disease. J Am Heart Assoc. 2016 Oct 12;5(10):e003807. doi: 10.1161/JAHA.116.003807. PMID 27733347
- [Derived] Mark DB, Federspiel JJ, Cowper PA, Anstrom KJ, Hoffmann U, Patel MR, Davidson-Ray L, Daniels MR, Cooper LS, Knight JD, Lee KL, Douglas PS; PROMISE Investigators. Economic Outcomes With Anatomical Versus Functional Diagnostic Testing for Coronary Artery Disease. Ann Intern Med. 2016 Jul 19;165(2):94-102. doi: 10.7326/M15-2639. Epub 2016 May 24. PMID 27214597
- [Derived] Mark DB, Anstrom KJ, Sheng S, Baloch KN, Daniels MR, Hoffmann U, Patel MR, Cooper LS, Lee KL, Douglas PS; PROMISE Investigators. Quality-of-Life Outcomes With Anatomic Versus Functional Diagnostic Testing Strategies in Symptomatic Patients With Suspected Coronary Artery Disease: Results From the PROMISE Randomized Trial. Circulation. 2016 May 24;133(21):1995-2007. doi: 10.1161/CIRCULATIONAHA.115.020259. Epub 2016 Apr 27. PMID 27143676
- [Derived] Douglas PS, Hoffmann U, Patel MR, Mark DB, Al-Khalidi HR, Cavanaugh B, Cole J, Dolor RJ, Fordyce CB, Huang M, Khan MA, Kosinski AS, Krucoff MW, Malhotra V, Picard MH, Udelson JE, Velazquez EJ, Yow E, Cooper LS, Lee KL; PROMISE Investigators. Outcomes of anatomical versus functional testing for coronary artery disease. N Engl J Med. 2015 Apr 2;372(14):1291-300. doi: 10.1056/NEJMoa1415516. Epub 2015 Mar 14. PMID 25773919
- [Derived] Douglas PS, Hoffmann U, Lee KL, Mark DB, Al-Khalidi HR, Anstrom K, Dolor RJ, Kosinski A, Krucoff MW, Mudrick DW, Patel MR, Picard MH, Udelson JE, Velazquez EJ, Cooper L; PROMISE investigators. PROspective Multicenter Imaging Study for Evaluation of chest pain: rationale and design of the PROMISE trial. Am Heart J. 2014 Jun;167(6):796-803.e1. doi: 10.1016/j.ahj.2014.03.003. Epub 2014 Mar 18. PMID 24890527

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Functional Diagnostic Tests | Anatomic Diagnostic Test
Started | 5007 | 4996
Completed | 3737 | 4123
Not Completed | 1270 | 873
Not completed — Death | 75 | 74
Not completed — Lost to Follow-up | 652 | 510
Not completed — Withdrawal by Subject | 543 | 289

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Functional Diagnostic Tests | Anatomic Diagnostic Test | Total
Number analyzed (Participants) | 5007 | 4996 | 10003
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (8.3) | 60.7 (8.3) | 60.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2675 | 2595 | 5270
  Male | 2332 | 2401 | 4733

OUTCOME MEASURES:

1. Primary Outcome: Time to Primary Endpoint
Description: Time to primary endpoint as defined as a composite of death, myocardial infarction (MI), major complications from cardiovascular (CV) procedures or testing, and unstable angina hospitalization. The Kaplan-Meier events rates (cumulative percentage of participants with an event) were estimated for the anatomic and functional diagnostic test groups.
Time Frame: 90 days, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months
Measure: Number; unit: Percentage of participants with an event
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 4996 | 5007
Percentage of participants with an event
  90 days | 1.0 | 1.1
  6 months | 1.2 | 1.4
  12 months | 1.8 | 1.9
  18 months | 2.5 | 2.6
  24 months | 2.9 | 2.8
  30 months | 3.5 | 3.5
  36 months | 4.6 | 3.8
  42 months | 5.3 | 5.1

2. Secondary Outcome: Time to Death, Myocardial Infarction (MI), Unstable Angina Hospitalization
Description: Time to this secondary endpoint as defined as a composite of death, myocardial infarction (MI), and unstable angina hospitalization. The Kaplan-Meier events rates (cumulative percentage of participants with an event) were estimated for the anatomic and functional diagnostic test groups.
Time Frame: 90 days, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months
Measure: Number; unit: Percentage of participants with an event
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 4996 | 5007
Percentage of participants with an event
  90 day | 0.9 | 1.0
  6 month | 1.2 | 1.4
  12 month | 1.8 | 1.9
  18 month | 2.5 | 2.5
  24 month | 2.9 | 2.8
  30 month | 3.5 | 3.4
  36 month | 4.6 | 3.7
  42 month | 5.2 | 5.1

3. Secondary Outcome: Time to Death or Myocardial Infarction (MI)
Description: Time to this secondary endpoint as defined as a composite of death and myocardial infarction (MI). The Kaplan-Meier events rates (cumulative percentage of participants with an event) were estimated for the anatomic and functional diagnostic test groups.
Time Frame: 90 days, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months
Measure: Number; unit: Percentage of participants with an event
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 4996 | 5007
Percentage of participants with an event
  90 Days | 0.3 | 0.6
  6 months | 0.4 | 0.9
  12 months | 0.8 | 1.2
  18 months | 1.3 | 1.8
  24 months | 1.7 | 2.0
  30 months | 2.2 | 2.7
  36 months | 3.3 | 3.0
  42 months | 3.9 | 4.2

4. Secondary Outcome: Time to Major Complications From Cardiovascular (CV) Procedures
Description: Time to this secondary endpoint as defined as a composite of major complications from cardiovascular procedures and testing (stroke, bleeding, anaphylaxis, renal failure). The Kaplan-Meier events rates (cumulative percentage of participants with an event) were estimated for the anatomic and functional diagnostic test groups.
Time Frame: 90 days, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months
Measure: Number; unit: Percentage of participants with an event
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 4996 | 5007
Percentage of participants with an event
  90 day | 0.1 | 0.3
  6 month | 0.2 | 0.5
  12 month | 0.5 | 0.8
  18 month | 1.0 | 1.1
  24 month | 1.2 | 1.4
  30 month | 1.7 | 1.9
  36 month | 2.6 | 2.2
  42 month | 3.1 | 3.2

5. Secondary Outcome: Time to Death, Myocardial Infarction (MI), Unstable Angina (UA), Complications, No Coronary Artery Disease (CAD)
Description: Time to primary endpoint as defined as a composite of death, myocardial infarction (MI), major complications from cardiovascular (CV) procedures or testing, unstable angina hospitalization, and no coronary artery disease (CAD). The Kaplan-Meier events rates (cumulative percentage of participants with an event) were estimated for the anatomic and functional diagnostic test groups.
Time Frame: 90 days, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months, 42 months
Measure: Number; unit: Percentage of participants with an event
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 4996 | 5007
Percentage of participants with an event
  90 days | 4.4 | 5.2
  6 months | 4.6 | 5.6
  12 months | 5.2 | 6.1
  18 months | 5.9 | 6.7
  24 months | 6.3 | 6.9
  30 months | 6.9 | 7.6
  36 months | 8.0 | 7.9
  42 months | 8.7 | 9.1

6. Secondary Outcome: Percentage of Invasive Cardiac Catheterization Events Without Obstructive Coronary Artery Disease Within 90 Days Following Participant Randomization
Description: Percentage of Invasive Cardiac Catheterization Events Without Obstructive Coronary Artery Disease (CAD)Within 90 Days Following Participant Randomization
Time Frame: Up to 90 days following participant randomization
Measure: Mean (Standard Error); unit: Percentage of events
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 4996 | 5007
Percentage of events | 3.4 (0.3) | 4.3 (0.3)

7. Secondary Outcome: Medical Cost
Description: Assess and compare total medical cost for the two diagnostic testing arms by intention to treat at both 90 days and 3 years cumulative.
Time Frame: 90 days and 3 years cumulative
Population: Patients enrolled in PROMISE and cared for in the fee-for-service sector of the US health care system were included in the economic study. Because the costing methods being used were not applicable to other health systems, patients enrolled in the Military/VA system , an Health maintenance Organization (HMO) , or in Canada were excluded.
Measure: Mean (95% Confidence Interval); unit: Per participant cost in US dollars
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 4818 | 4831
Per participant cost in US dollars
  90 days | 2494 [2233 to 2821] | 2240 [1599 to 3119]
  3 years cumulative | 7213 [6501 to 8156] | 6586 [5683 to 7772]

8. Secondary Outcome: Quality of Life (QOL) as Measured by Duke Activity Status Index
Description: Participant score in Quality of Life as measured by Duke Activity Status Index (DASI). DASI measures a person's functional capacity based on a 12-item questionnaire that correlates with peak O2 uptake during exercise testing. The DASI is a self-administered questionnaire that measures a patient's functional capacity. It can be used to get a rough estimate of a patient's peak oxygen uptake. The maximum score for the DASI is 58.2 (better functional ability/capacity) and the minimum score is 0 (worse functional ability/capacity).
Time Frame: Baseline, 6 months, 12 months 24 months
Population: The number of participants were limited due to budget constraints.
Measure: Median (Inter-Quartile Range); unit: participant score
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 2982 | 3003
participant score
  Baseline | 21.5 [10.7 to 38.2] | 22.9 [10.0 to 39.5]
  6 months | 30.5 [10.7 to 44.7] | 30.2 [15.2 to 44.7]
  12 months | 29.2 [13.5 to 44.7] | 31.2 [15.2 to 44.7]
  24 months | 31.5 [16.0 to 45.5] | 31.2 [16.0 to 45.5]

9. Secondary Outcome: Quality of Life (QOL) as Measured by Seattle Angina Scale Anginal Frequency Subscale
Description: Participant score Quality of Life measured by Seattle Angina Scale Anginal Frequency Subscale utilizing the Seattle Angina Questionnaire (SAQ). SAQ: 19-item, 5-6-point Likert, questionnaire measuring 5 dimensions of coronary artery disease: Anginal Stability: whether symptoms are changing. Anginal Frequency: how often patient having symptoms Physical Limitation: how much condition hampers ability to do what he wants.Treatment Satisfaction: how well patient understands care. Disease Perception: impact of condition on interpersonal relationships. Each dimension assigns response an value, beginning with 1 for response at the lowest level of functioning & summing across items within each of the 5 scales. Scale scores transformed to 0-100 range by subtracting the lowest scale. Higher score suggest symptoms more stable & less frequent, condition has less impact on activities, increased satisfaction with treatment, & perception of disease has less impact on interpersonal relationships.
Time Frame: Baseline, 6 month, 12 month, 24 month
Population: The number of participants were limited due to budget constraints.
Measure: Median (Inter-Quartile Range); unit: participant score
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 2982 | 3003
participant score
  Baseline | 70 [70 to 90] | 80 [70 to 90]
  6 month | 100 [90 to 100] | 100 [90 to 100]
  12 month | 100 [90 to 100] | 100 [90 to 100]
  24 month | 100 [100 to 100] | 100 [100 to 100]

10. Secondary Outcome: Quality of Life (QOL) as Measured by Seattle Anginal Quality of Life Subscale
Description: as for outcome 9
Time Frame: Baseline, 6 months, 12 months, 24 months
Population: The number of participants were limited due to budget constraints.
Measure: Median (Inter-Quartile Range); unit: participant score
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 2982 | 3003
participant score
  Baseline | 58.3 [41.7 to 75.0] | 58.3 [41.7 to 75.0]
  6 month | 83.3 [75.0 to 91.7] | 83.3 [75.0 to 100]
  12 month | 83.3 [75.0 to 100] | 91.7 [75.0 to 100]
  24 month | 91.7 [75 to 100] | 91.7 [75.0 to 100]

11. Secondary Outcome: Quality of Life (QOL) as Measured by Complete Resolution of Symptoms That Led to the Initial Testing
Description: Percentage of participants with improvement in Quality of Life as measured by complete resolution of the symptoms that led to initial testing
Time Frame: 6 month, 12 month 24 month
Population: The number of participants were limited due to budget constraints.
Measure: Number; unit: % of participants
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 2982 | 3003
% of participants
  6 months | 43.3 | 46.5
  12 months | 47.3 | 48.8
  24 months | 52.1 | 54.3

12. Secondary Outcome: Cumulative Radiation Exposure Within 90 Days
Description: Cumulative radiation exposure from all cardiovascular diagnostic tests and procedures performed within 90 days after randomization.
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: milliSievert (mSv)
Arm/Group | Anatomic Diagnostic Test | Functional Diagnostic Tests
Number analyzed (Participants) | 4996 | 5007
milliSievert (mSv) | 10.0 [5.6 to 17.2] | 11.3 [0.0 to 13.5]

ADVERSE EVENTS:
Time Frame: Events occuring within 24 hours following the study intervention (initial test) were collected and reported by study personnel.
Description: Severe Events/complications related to cardiovascular testing or cardiovascular procedures that are trial endpoints were collected throughout the duration of the trial and were considered related to testing or procedure only if occuring within 72 hours of test or procedure.
Arm/Group | Functional Diagnostic Tests | Anatomic Diagnostic Test
Serious Adverse Events (participants affected / at risk) | 161/5007 | 168/4996
Other Adverse Events (participants affected / at risk) | 16/5007 | 37/4996
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Functional Diagnostic Tests (N=5007) | Anatomic Diagnostic Test (N=4996)
Death- Cardiovascular (Cardiac disorders) | 21 | 14
Major Bleeding (Cardiac disorders) | 3 | 3
Myocardial Infarction (Cardiac disorders) | 40 | 30
Stroke (Cardiac disorders) | 2 | 1
Unstable Angina Hospitalization (Cardiac disorders) | 41 | 61
Death - Non cardiovascular known cause (General disorders) | 27 | 33
Death - unknown cause (General disorders) | 27 | 27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Functional Diagnostic Tests (N=5007) | Anatomic Diagnostic Test (N=4996)
Exercise Induced Hypotension (Cardiac disorders) | 6 | 0
Stress Induced Symptoms Related to Functional Testing (Cardiac disorders) | 4 | 0
Ventricular Tachycardia (Cardiac disorders) | 4 | 0
Hemodynamic Instability (Cardiac disorders) | 2 | 3
Hospital Admission Not In The Primary Endpoint (General disorders) | 5 | 0
Any Event Potentially Related to Vasodilators (Cardiac disorders) | 5 | 0
Mild Contrast Reaction (rash or hives) (Skin and subcutaneous tissue disorders) | 0 | 22
Extravasion of Contrast Into Surrounding Tissue (Skin and subcutaneous tissue disorders) | 0 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No